CLINICAL TRIAL: NCT04032262
Title: Characterization of Gastrointestinal and Neuroenteric Dysfunction in Parkinson's Disease
Brief Title: Parkinson's Disease and Digestive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Parkinson's Disease Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PARKIDF00001
Record Dates: First submitted 2018-04-19; First posted 2019-07-25 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Constipation; Gastro-Intestinal Disorder
Keywords: Brain-Gut Relationship; Anorectal Manometry
MeSH Terms: conditions — Parkinson Disease; Constipation; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Parkinson's Disease Relationship to the GI track (Other): Patients with Parkinson's.
  Interventions: Diagnostic Test: Gastrointestinal and Parkinson's Disease

INTERVENTIONS:
Diagnostic Test: Gastrointestinal and Parkinson's Disease — Subjects with Parkinson's disease will come for visits that will contain questionnaires about their PD, their bowel movements, and do further tests using anal rectal probes to understand further their constipation, and other tests to gather data on their digestion.

SUMMARY:
This study focuses on the relationship between the brain and the gut, and additionally will foster collaboration between Movement Disorder experts and Neurogastroenterologists to provide critical information and lead to innovative therapies in the future to treat GI dysfunction of Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's disease affects 1 million people in the US with a rising prevalence. In addition to neurological problems, patients with Parkinson's Disease often suffer from debilitating gastrointestinal (GI) symptoms related to delayed stomach emptying, gas/bloating, and constipation. GI complaints of patients suffering from Parkinson's Disease are poorly understood. This proposal aims to characterize GI disturbance in patients with Parkinson's Disease and provide deeper understanding by investigating symptoms, regional and whole gut transit, anorectal physiology, and the brain-gut axis. The investigator believes patients with Parkinson's Disease will show altered GI sensation, slower GI motility and demonstrate deranged regulation of the brain-gut axis correlated to severity of Parkinson's disease. Results from this study of GI motility and brain-gut axis will define a subset of Parkinson's Disease patients that can benefit from tailored treatment. This study will foster collaboration between Movement Disorder experts and Neurogastroenterologists to provide critical information and lead to innovative therapies in the future to treat GI dysfunction of Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Presence of 2 of 3 cardinal features of PD (resting tremor, bradykinesia, and rigidity)
* Hoehn and Yahr Scale stage I-IV
* Men or women aged 18+
* Stable dopaminergic treatment for ≥4 weeks.
* Women of childbearing potential must agree to a urine pregnancy test at screening and to avoid pregnancy throughout the study.

Exclusion Criteria:

* Secondary parkinsonism.
* Parkinson-plus syndromes.
* Montreal Cognitive Assessment score <17.
* Unstable dosage of drugs active in the cns (e.g., anxiolytics, antidepressants) during the 60 days before the visit.
* Participation in drug studies within 30 days of screening.
* Structural brain disease.
* Women who are pregnant or likely to conceive (women with potential for pregnancy must use contraceptive measures to be included);
* Active or personal history of epilepsy.
* Acute illness or active, confounding medical, neurologic, or musculoskeletal conditions.
* Alcoholism or other forms of drug addiction.
* Significant prior gastrointestinal surgery.
* Ongoing chemotherapy or other treatment for cancer.
* Dysphagia
* implanted or externally worn medical device such as, but not limited to, a pacemaker. (gastric stimulators, bladder stimulators, spinal stimulators, medication infusion devices, insulin pumps, continuous glucose monitors are permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Cortical Evoked Potential (CEP) | Single Visit, 3 hours
  Bilateral amplitude (microvolts) for ano-rectal CEP responses
Motor Evoked Potential (MEP) | Single visit, 2 hours
  Bilateral amplitude (microvolts) for ano-rectal MEP responses

SECONDARY OUTCOMES:
Gastrointestinal motor function and transit | 2 visits, 1hour
  The measurements to be obtained are gastric emptying time (GET), small bowel transit time (SBTT), colonic transit time (CTT) and whole gut transit time (WGTT) over a period of 5 days. Tool to be used includes wireless motility capsule and corresponding recorder swallowed on initial visit and returned 5 days later. Specific measurements obtained include time in hours of GET, SBTT, CTT, WGTT. These outcome will only be measured once per subject and not be reassessed.
Rectal sensorimotor function | Single visit, 2 hours
  Rectal sustained squeeze pressure (mmHg) measure from Anal rectal manometry study
Anal sensorimotor function | Single visit, 2 hours
  Anal sustained squeeze pressure (mmHg) measure from Anal rectal manometry study
Unified Parkinson Disease Rating Scale (UPDRS) | Single visit, 1 hour
  Used to follow the longitudinal course of Parkinson's disease. The UPDRS scale consists of the following five segments: 1) Mentation, Behavior, and Mood, 2) ADL, 3) Motor sections, 4) Modified Hoehn and Yahr Scale, and 5) Schwab and England ADL scale. Some sections of the UPDRS scale require multiple grades assigned to each extremity with a possible maximum of 199 points. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).
Montreal Cognitive Assessment (MoCA) | Single visit, 1 hour
  Screening assessment for detecting cognitive impairment. MoCA scores range between 0 and 30. A final total score of 26 and above is considered normal.
Non-motor symptoms questionnaire | Single visit, 1 hour
  A 30-item screening patient-based questionnaire used to determine the non-motor symptoms experienced by the patient. The points should be totalled to give a score out of 30. A score of under 10 is mild, 10-20 moderate and over 20, severe.
36-Item Short Form Survey (SF-36) | Single visit, 1 hour
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Stool diary | 2 visits, 1 hour
  The measurement to be obtained is bowel pattern. Tool to be used include 2-week stool diary. Specific measurements obtained include number of complete spontaneous bowel movements (CSBMs) a week. These outcome will only be measured once per subject and not be reassessed.
Gastroparesis Cardinal Symptom Index (GCSI) | Single visit, 1 hour
  The GCSI is based on three subscales: post-prandial fullness/early satiety (4 items); nausea/vomiting (3 items), and bloating (2 items). A six-point Likert response scale, ranging from 0 (none) to 5 (very severe), with a 2-week recall period, was used to rate the severity of each symptom. The GCSI total score was constructed as the average of the three symptom sub-scales. GCSI total scores were in the range 0-5, with higher scores reflecting greater symptom severity.
Eckdart score (ESS) | Single visit, 1 hour
  The ESS is a 4 item self-report scale measuring weight loss in kilograms, chest pain, regurgitation, and dysphagia. Each item is graded on a score of 0 to 3, with a maximum score of 12. Scores greater than or equal to 3 are considered suggestive of active achalasia. The ESS is widely used in both clinical and research settings as a gold standard for measuring achalasia symptom severity.
Breath testing | Single visit, 3 hours
  The measurement to be obtained is presence of bacterial overgrowth. Tool to be used include breath testing via gas chromatography. Specific measurements obtained hydrogen and methane in parts per million (ppm) at baseline and every 30 minutes for 2-3 hours. These outcome will only be measured once per subject and not be reassessed.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Sharma, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University Digestive Health Research, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Parkinson's Disease foundation sponsored this study they will most likely be made aware about how recruitment went, participation, and ending results.